CLINICAL TRIAL: NCT05538013
Title: Investigation of the Relationship of Obesity Awareness With Physical Activity Level and Sedentary Behavior in Obese Women
Brief Title: Obesity Awareness, Physical Activity Level and Sedentary Behavior in Obese Women
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc. Prof., Biruni University
Other Study IDs: 2022/71-12
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Obesity
Keywords: obesity; women; physical activity; sedantary
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obese women: The study will consist of 70 obese women volunteers aged between 18-65 years.
  Interventions: Other: Survey evaluation

INTERVENTIONS:
Other: Survey evaluation — Obesity awareness, physical activity, and sedentary time questionnaires will be applied to these cases.

SUMMARY:
It is known that the incidence of obesity, which is a global health problem, is higher in women. The aim of this study is to examine the relationship of obesity awareness with physical activity level and sedentary behavior in obese women.

DETAILED DESCRIPTION:
Obese people are at risk for medical conditions that can lead to greater morbidity and mortality. It is known that the incidence of obesity, which is a global health problem, is higher in women. Lack of physical activity and sedentary behavior are well-known risk factors for obesity and the relationship between them has been supported by many studies. As a matter of fact, some studies have reported that public health programs should focus on increasing individuals' physical activity levels as well as reducing sitting time. While examining the sedentary behavior and physical activity levels of obese women, evaluating their obesity awareness status, can facilitate increasing their awareness of the disease, initiating and complying with treatment. The aim of this study is to examine the relationship of obesity awareness with physical activity level and sedentary behavior in obese women.

ELIGIBILITY:
Inclusion Criteria:

* The women who are ages between 18-65 years,
* BMI ≥ 30.0 kg/m2 according to WHO classification.

Exclusion Criteria:

* BMI < 30.0 kg/m2 according to WHO classification,
* Male participants,
* Inability to cooperate with assessments,
* Those who have had severe trauma or surgery that limit physical activities in the last 6 months,
* Those who have orthopedic, neurological, cardiovascular problems that limit / prevent ambulation,
* Pregnancy or suspected pregnancy,
* Individuals are included in a rehabilitation program.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will consist of 70 obese women volunteers aged between 18-65 years.
Study Population: The study will consist of 70 obese women volunteers aged between 18-65 years.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Obesity Awareness | baseline
  Obesity awareness will be measured by Obesity Awareness Insight Scale and Obesity.

SECONDARY OUTCOMES:
Sedentary Behavior Questionnaire | baseline
  It is a questionnaire developed to evaluate the time spent performing 9 sedentary behaviors on a normal weekday and weekend day. The questionnaire has nine different response options. For the total score, the durations of the behaviors in hours are added separately as weekdays and weekends. To obtain the average sedentary behavior times for weekdays and weekends, the total duration of the week is multiplied by 5, and the total duration of the weekend is multiplied by 2.
International Physical Activity Questionnaire Short Form | baseline
  The questionnaire allows calculation of metabolic equivalent (MET) by measuring frequency, duration and physical activity intensity level in the last seven days and shows weekly physical activity amount. It is calculated as weekly working hours (MET-min/week). Physical activity levels of individuals according to the calculated MET value: (1) <600 MET-min/week not active (sedentary, inactive), (2) 600-3000 MET-min/week minimally active, and (3) >3000 MET-min/week very active (physical activity that increases well-being) classified as.
Waist circumference | baseline
  Waist circumference will be measured with a tape measure in the standing position, by determining the midpoint between the lowest rib and the iliac crest from the exposed waist circumference.
Body fat-muscle ratios | baseline
  These measurements will be determined by bioelectrical impedance.

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, PT, PhD, Study Chair — Biruni University
Locations (1):
- Bezmi Alem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If the journal asks for the data, we will share it.